CLINICAL TRIAL: NCT03429309
Title: The Association Between Telomere Length in Peripheral Blood Leukocyte and Propofol Dose in Anesthesia-induction
Brief Title: The Association Between Telomere Length and Propofol Dose in Anesthesia-induction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guangzhou General Hospital of Guangzhou Military Command (Other)
Responsible Party: Principal Investigator, Weifeng Tu, Chief physician, Guangzhou General Hospital of Guangzhou Military Command
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Telomere length and propofol
Record Dates: First submitted 2017-11-21; First posted 2018-02-12 (Actual); Last update posted 2018-02-12 (Actual); Status verified 2017-11

CONDITIONS: General Anesthesia
Keywords: telomere; propofol; anesthesia-induction
MeSH Terms: interventions — Propofol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Anesthesia-induction with propofol (Other)
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Propofol — Anesthesia was induced by intravenous infusion of propofol via the syringe pump at a rate of 30 mg/kg/h.

SUMMARY:
Telomeres are protein-bound DNA repeat structures at the end of eukaryotic chromosomes that are made up of a simple repetitive sequence (in humans, TTAGGG) and regulate cellular replicative capacity and cellular proliferation, protect chromosomes from fusing together during mitosis and maintain genomic stability, and prevent the loss of genetic data. Telomeres are specialized repetitive DNA sequences, typically ranging from 5,000 to 15,000 bp in humans, which are the critical chromosome capping DNA sequences. The loss of telomere repeats diminishes telomeric functional capacity.Telomere length(TL) is important in determining telomere function.This is known as the end replication problem and results in a gradual decline in TL over time. Consequently,leukocyte TL shortens in a predictable way with age by roughly 20-40 base pairs per year. Cellular senescence and subsequent cell death often occur when the mean telomere length reaches a critical value.Shortened telomeres and lower telomerase are linked to age-related risk factors and disease.Peripheral blood leukocyte express telomerase at low levels, which can be measured over a short duration (hours) to demonstrate immediate, short-term changes. Shorter mean leukocyte telomere length has been shown to be associated with risk of several age-related diseases.The dosage of propofol gradually reduced with the aging process. However,it is not known whether the telomere length and variation of telomerase in PBL relate to the dosage of propofol and time of consciousness disappearance in anesthesia induction. In this exploratory study, the investigators examined that the changes of peripheral blood leukocyte telomere length was associated with the dosage of propofol and time of consciousness disappearance in anesthesia induction.

Given the importance of telomeres in nuclear and cellular function, the central role of telomere length in determining telomere function,the investigator study that the changes of telomere length in peripheral blood leukocyte of patients are associated with the dosage of propofol in anesthesia induction.

DETAILED DESCRIPTION:
A hundred patients with the American Society of Anesthesiologists (ASA) physical status I-II, aged from 18 to 80 years, gave an informed-written consent to participate.Testing took place in the morning after an overnight fast. Patients were scheduled for elective surgical procedures. After arrival to the operating theater, the peripheral venous line for fluid and drug administration was inserted. The electrocardiogram, heart rate, a noninvasive blood pressure, a pulse oximeter and bispectral (BIS) Index were monitored continuously. 100% oxygen was given for 3 min by face mask. Anesthesia was induced by intravenous infusion of propofol via the syringe pump at a rate of 30 mg/kg/h. Recordings began before propofol induction started. After the start of the propofol infusion and BIS Index at 80, patients were asked loudly "open eyes" and examined eyelash reflex at 15-s intervals until loss of consciousness (unresponsiveness to the verbal command, no spontaneous movements and loss of eyelash reflex); and recordings of the heart rate, a noninvasive blood pressure and BIS Index were obtained during awake baseline and unconsciousness induced by propofol. Propofol dosage and consciousness disappearance time were recorded after propofol-induced loss of consciousness. The commands were spoken in a loud voice by the investigator and were repeated up to three times, if the subject failed to respond. A subject who obeyed command was considered conscious. The BIS index is useful, and a reliable and sensitive indicator for assessing the level of consciousness during sedation and hypnosis with propofol so that the investigators recorded BIS index to evaluate level of consciousness. To minimize artifacts, patients were instructed not to open their eyes, talk, or move during the heart rate, a noninvasive blood pressure and BIS Index recordings before the propofol infusion and the sedation level was assessed until the patient's unconsciousness.

ELIGIBILITY:
Inclusion Criteria:

* Patients were scheduled for elective surgical procedures

Exclusion Criteria:

* patients with known cardiac, pulmonary, renal disease, hearing disorders or neurological diseases, diabetes, and patients taking drugs affecting to the central nervous system or consuming more than 20 g alcohol daily, a body mass index>30

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-12-01 (Actual); Primary Completion 2018-02-01 (Actual); Study Completion 2018-02-28 (Estimated)

PRIMARY OUTCOMES:
Propofol Dose | through study completion, up to 6 months
  Dosage of propofol in anesthesia-induction.
Telomere Length | through study completion, up to 6 months
  Telomere length of peripheral blood leukocyte

SECONDARY OUTCOMES:
Time of anesthesia-induction. | through study completion, up to 6 months
  Time counted from the beginning of anesthesia-induction to patient consciousness disappearance.
HR | through study completion, up to 6 months
  Heart Rate
BP | through study completion, up to 6 months
  Blood Pressure
BIS | through study completion, up to 6 months
  BIS index

CONTACTS AND LOCATIONS:
Locations (1):
- Guangzhou General Hospital of Guangzhou Military Command, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Blackburn EH, Greider CW, Szostak JW. Telomeres and telomerase: the path from maize, Tetrahymena and yeast to human cancer and aging. Nat Med. 2006 Oct;12(10):1133-8. doi: 10.1038/nm1006-1133. No abstract available. PMID 17024208
- [Background] Aubert G, Lansdorp PM. Telomeres and aging. Physiol Rev. 2008 Apr;88(2):557-79. doi: 10.1152/physrev.00026.2007. PMID 18391173
- [Background] Biegler KA, Anderson AK, Wenzel LB, Osann K, Nelson EL. Longitudinal change in telomere length and the chronic stress response in a randomized pilot biobehavioral clinical study: implications for cancer prevention. Cancer Prev Res (Phila). 2012 Oct;5(10):1173-82. doi: 10.1158/1940-6207.CAPR-12-0008. Epub 2012 Jul 24. PMID 22827974
- [Background] Starkweather AR, Alhaeeri AA, Montpetit A, Brumelle J, Filler K, Montpetit M, Mohanraj L, Lyon DE, Jackson-Cook CK. An integrative review of factors associated with telomere length and implications for biobehavioral research. Nurs Res. 2014 Jan-Feb;63(1):36-50. doi: 10.1097/NNR.0000000000000009. PMID 24335912
- [Background] Munoz P, Blanco R, Blasco MA. Role of the TRF2 telomeric protein in cancer and ageing. Cell Cycle. 2006 Apr;5(7):718-21. doi: 10.4161/cc.5.7.2636. Epub 2006 Apr 1. PMID 16582635
- [Background] Codd V, Mangino M, van der Harst P, Braund PS, Kaiser M, Beveridge AJ, Rafelt S, Moore J, Nelson C, Soranzo N, Zhai G, Valdes AM, Blackburn H, Mateo Leach I, de Boer RA, Kimura M, Aviv A; Wellcome Trust Case Control Consortium; Goodall AH, Ouwehand W, van Veldhuisen DJ, van Gilst WH, Navis G, Burton PR, Tobin MD, Hall AS, Thompson JR, Spector T, Samani NJ. Common variants near TERC are associated with mean telomere length. Nat Genet. 2010 Mar;42(3):197-9. doi: 10.1038/ng.532. Epub 2010 Feb 7. PMID 20139977
- [Background] Cesare AJ, Reddel RR. Alternative lengthening of telomeres: models, mechanisms and implications. Nat Rev Genet. 2010 May;11(5):319-30. doi: 10.1038/nrg2763. Epub 2010 Mar 30. PMID 20351727
- [Background] Capezzone M, Cantara S, Marchisotta S, Filetti S, De Santi MM, Rossi B, Ronga G, Durante C, Pacini F. Short telomeres, telomerase reverse transcriptase gene amplification, and increased telomerase activity in the blood of familial papillary thyroid cancer patients. J Clin Endocrinol Metab. 2008 Oct;93(10):3950-7. doi: 10.1210/jc.2008-0372. Epub 2008 Jul 29. PMID 18664542
- [Background] Epel ES, Lin J, Dhabhar FS, Wolkowitz OM, Puterman E, Karan L, Blackburn EH. Dynamics of telomerase activity in response to acute psychological stress. Brain Behav Immun. 2010 May;24(4):531-9. doi: 10.1016/j.bbi.2009.11.018. Epub 2009 Dec 16. PMID 20018236
- [Background] Humphreys J, Epel ES, Cooper BA, Lin J, Blackburn EH, Lee KA. Telomere shortening in formerly abused and never abused women. Biol Res Nurs. 2012 Apr;14(2):115-23. doi: 10.1177/1099800411398479. Epub 2011 Mar 8. PMID 21385798